CLINICAL TRIAL: NCT05289063
Title: Vascular Endothelial Dysfunction in Sleep Apnea
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sanja Jelic, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AAAT8810; 2R01HL106041 (NIH)
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: CPAP; Atorvastatin
MeSH Terms: interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Intervention Model Description: Randomized double blind design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active drug and placebo will be made identical in appearance and given to participants in a blinded fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): OSA patients who adhered or did not adhere with CPAP who are randomized to receive atorvastatin 10 mg daily.
  Interventions: Drug: Atorvastatin 10mg; Other: Continuous Positive Airway Pressure Therapy
- Control (Placebo Comparator): OSA patients who adhered or did not adhere with CPAP who are randomized to receive placebo daily.
  Interventions: Drug: Placebo; Other: Continuous Positive Airway Pressure Therapy

INTERVENTIONS:
Drug: Atorvastatin 10mg — Atorvastatin 10 mg daily for 28 days will be randomly allocated to OSA patients regardless of adherence with CPAP. Atorvastatin and placebo will be encapsulated to appear identical and dispensed by the research pharmacy.
  Other Names: statin
  Arms: Treatment
Drug: Placebo — Placebo daily for 28 days will be randomly allocated to OSA patients regardless of adherence with CPAP. Atorvastatin and placebo will be encapsulated to appear identical and dispensed by the research pharmacy.
  Arms: Control
Other: Continuous Positive Airway Pressure Therapy — CPAP is a standard of care for OSA and will be prescribed by care providers not associated with this study based on clinical indications. The investigators will have no role in prescribing CPAP.
  Other Names: CPAP

SUMMARY:
This double-blind placebo-controlled parallel group randomized study design will be used to test whether 4 weeks of atorvastatin 10 mg daily reduces levels of inflammatory markers in OSA patients treated with CPAP (standard of care). The purpose of this study is to investigate: 1) whether statins reduce endothelial inflammation and pro-thrombotic conditions in OSA, including in patients adherent to CPAP (Aim 1); and 2) whether statins reduce endothelial inflammation and pro-thrombotic conditions by improving endothelial cholesterol metabolism and trafficking in OSA (Aim 2).

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA), a condition that affects a quarter of American adults, triples the risk for cardiovascular diseases and increases all-cause mortality. Standard therapy with continuous positive airway pressure (CPAP) does not improve cardiovascular risk. Based on the investigators' mechanistic observation that the abnormal cycle of endothelial inflammation can be disrupted with statin therapy, the investigators now propose randomized clinical trial of statins vs. placebo to determine its effects on endothelial dysfunction in OSA patients treated with CPAP, which may provide the basis for practical clinical trials of statins for reducing cardiovascular risk in OSA.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Newly diagnosed with obstructive sleep apnea (OSA) who were never treated with CPAP. OSA is defined as apnea-hypopnea index (AHI) ≥5 events/hour of sleep.

Exclusion Criteria:

* A history of coronary artery disease, heart failure, stroke, diabetes, malignancy, chronic pulmonary, kidney or rheumatologic disease, muscle pain/fatigue, smoking within the past 5 years
* Regular use of any medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Circulating levels of Angiopoietin-2 after 4 weeks of atorvastatin vs. placebo therapy | 4 weeks post-treatment
  Mean circulating levels of Ang-2 will be quantified after 4 weeks of statin or placebo therapy by enzyme-linked immunosorbent assay (ELISA)
Interaction of endoplasmic reticulum (ER)-bound vesicle-associated membrane protein-associated protein B (VAPB) with late endosome-bound ORP1L (proximity ligation assay fluorescence area in µm2) after 4 weeks of atorvastatin vs. placebo therapy | 4 weeks post-treatment
  Mean Interactions ER-bound VAPB with late endosome-bound ORP1L in harvested endothelial cells (ECs) will be assessed using proximity ligation assay (DuoLink, fluorescence area in µm2) after 4 weeks of atorvastatin or placebo therapy

SECONDARY OUTCOMES:
Circulating levels of von Willebrand factor cleavage products after 4 weeks of atorvastatin vs. placebo | 4 weeks post-treatment
  Mean Circulating levels (count) of von Willebrand factor (vWF) cleavage products (low molecular weight (LMW), medium molecular weight (IMW), high molecular weight (HMW)) after 4 weeks of atorvastatin vs. placebo
Circulating levels of von Willebrand factor (vWF) cleavage products (low, medium, high molecular weight) at baseline and after 4 weeks of CPAP | 4 weeks post-CPAP
  Mean Circulating levels (count) of vWF cleavage products (LMW, IMW, HMW) at baseline and after CPAP.
Endothelial cell free cholesterol levels after 4 weeks of atorvastatin vs. placebo | 4 weeks post-treatment
  Mean Endothelial cell free cholesterol levels (fluorescence intensity) after 4 weeks of atorvastatin vs. placebo therapy
Endothelial cell lipid droplets after 4 weeks of atorvastatin vs. placebo | 4 weeks post-treatment
  Mean Endothelial cell lipid droplets (fluorescence area µm2) after 4 weeks of atorvastatin vs. placebo
Endothelial cell interactions between CD59 and Weibel Palade Bodies (WPBs) after 4 weeks of atorvastatin vs. placebo | 4 weeks post-treatment
  Mean Endothelial cell interactions between CD59 and Weibel Palade Bodies (fluorescence area µm2) after 4 weeks of atorvastatin vs. placebo
Circulating levels of Angiopoietin-2 at baseline and after 4 weeks of CPAP therapy | 4 weeks post-CPAP
  Mean Circulating levels of Angiopoietin-2 after 4 weeks of CPAP therapy quantified by ELISA
Interaction of ER-bound VAPB with late endosome-bound ORP1L (proximity ligation assay fluorescence area in µm2) at baseline and after 4 weeks of CPAP therapy | 4 weeks post-CPAP
  Mean Interaction of ER-bound VAPB with late endosome-bound ORP1L (proximity ligation assay fluorescence area in µm2) after 4 weeks of CPAP therapy
Endothelial cell nuclear factor kappa B (NF-κB) nuclear fluorescence intensity after 4 weeks of atorvastatin vs. placebo | 4 weeks post-treatment
  Mean Endothelial cell NF-kB nuclear fluorescence intensity after 4 weeks of atorvastatin vs. placebo
Circulating levels of E-selectin after 4 weeks of atorvastatin vs. placebo therapy | 4 weeks post-treatment
  Mean Circulating levels of E-selectin after 4 weeks of atorvastatin vs. placebo therapy quantified by ELISA
Endothelial cell messenger ribonucleic acid (mRNA) expression of EC adhesion molecules after 4 weeks of atorvastatin vs. placebo | 4 weeks post-treatment
  Mean Endothelial cell mRNA expression of EC adhesion molecules after 4 weeks of atorvastatin vs. placebo quantified by reverse transcription polymerase chain reaction (RT-PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Sanja Jelic, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No